CLINICAL TRIAL: NCT02081248
Title: Easy-to-Read Informed Consent (ETRIC) for Hematopoietic Cell Transplantation Clinical Trials (BMT CTN #1205)
Brief Title: Easy-to-Read Informed Consent (ETRIC) for Hematopoietic Cell Transplantation Clinical Trials (BMT CTN 1205)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BMTCTN1205; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2013-10-30; First posted 2014-03-07 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Improve the Informed Consent Process

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Consent (Active Comparator): This arm will receive the Consent Form Specific Format 1 'standard consent'. The standard consents are already approved and used for the BMT CTN 0901, 1101, 1203, and 1301 trials.
  Interventions: Other: Consent Form Specific Format 1
- Easy-to-Read Informed Consent (Experimental): This arm will receive the Consent Form Specific Format 2 'Easy-to-Read Informed Consent'.The Easy-to-Read Informed Consent (ETRIC) is the newly approved consent.
  Interventions: Other: Consent Form Specific Format 2

INTERVENTIONS:
Other: Consent Form Specific Format 1 — The Consent Form Specific Format 1 is the 'Standard Consent'. The standard consent does not have the format of two-columns with changes in layout readability, organization of content, typography and use of plain language. Standard consents are already used by sites for the BMT CTN 0901, 1101, 1203, and 1301 clinical trials.
  Arms: Standard Consent
Other: Consent Form Specific Format 2 — The Consent Form Specific Format 2 is the 'Easy-to-Read Informed Consent'.The Easy-to-Read Informed Consent is two-columns with changes in layout readability, organization of content, typography and use of plain language.
  Arms: Easy-to-Read Informed Consent

SUMMARY:
The study has two parts: (1) Randomized Study to evaluate the effectiveness of ETRIC, and (2) Evaluation Study to understand barriers to implementation of ETRIC.

DETAILED DESCRIPTION:
A two-arm, randomized study will be conducted in patients about to undergo consent discussion for participation in two large, multicenter BMT CTN clinical trials. Once they agree to participate in this Easy-to-Read Informed Consent (ETRIC) study, they will go through the consent process for the parent trial using either a standard or the ETRIC consent form. The content of both forms will be similar but the ETRIC form will incorporate a two-column format with specific attention towards enhanced readability and processability. Following the consent discussion for the BMT CTN parent trial, patients will complete assessments of health literacy, comprehension of the parent trial and satisfaction and anxiety related to the consent process. These assessments will be completed within 7 business days of the consent discussion of the parent trial.

Notes: Enrollment on the BMT CTN 0901 trial (NCT01339910) was closed to further accrual on April 18, 2014. Enrollment on the BMT CTN 1203 trial (NCT02208037) completed accrual on May 13, 2016.

ELIGIBILITY:
Inclusion and exclusion criteria for the ETRIC randomized study will be the same as the eligibility criteria for the BMT CTN parent studies. Please refer to BMTCTN0901 (NCT01339910) Reduced Intensity Regimen vs Myeloablative Regimen for Myeloid Leukemia or Myelodysplastic Syndrome, BMTCTN1101 (NCT01597778) Double Cord Versus Haploidentical, BMTCTN1203 (NCT02208037) Novel Approaches for Graft-versus-Host Disease Prevention Compared to Contemporary Controls, and BMTCTN1301 (NCT02345850) Calcineurin Inhibitor-Free Interventions for Prevention of Graft-versus-Host Disease for detailed eligibility criteria.

Notes: Enrollment on the BMT CTN 0901 trial (NCT01339910) was closed to further accrual on April 18, 2014. Enrollment on the BMT CTN 1203 trial (NCT02208037) completed accrual on May 13, 2016.

Additional inclusion criteria specific for the ETRIC study will include:

1. Adult patients (≥ 18 years)
2. Speaking and reading proficiency in English (as most of this study's instruments have not been translated and validated in languages other than English)
3. Willing and able to provide informed consent
4. Stated willingness to comply with study procedures and reporting requirements

Exclusion Criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (23):
- United States (23):
  - City of Hope National Medical Center, Duarte, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - BMT Program at Northside Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas, Lawrence, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - West Virginia University Hospital, Morgantown, West Virginia
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript.
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Spellecy R, Tarima S, Denzen E, Moore H, Abhyankar S, Dawson P, Foley A, Gersten I, Horwitz M, Idossa L, Joffe S, Kamani N, King R, Lazaryan A, Morris L, Horowitz MM, Majhail NS. Easy-to-Read Informed Consent Form for Hematopoietic Cell Transplantation Clinical Trials: Results from the Blood and Marrow Transplant Clinical Trials Network 1205 Study. Biol Blood Marrow Transplant. 2018 Oct;24(10):2145-2151. doi: 10.1016/j.bbmt.2018.04.014. Epub 2018 Apr 18. PMID 29679770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Started | 98 | 100
Completed | 76 | 87
Not Completed | 22 | 13

BASELINE CHARACTERISTICS:
Population: Enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Consent | Easy-to-Read Informed Consent | Total
Number analyzed (Participants) | 98 | 100 | 198
Age, Continuous [Median (Full Range); unit: years] | 61 [27 to 73] | 61 [21 to 76] | 61 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 53 | 57 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 87 | 94 | 181
  Unknown or Not Reported | 6 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 85 | 88 | 173
  Black | 7 | 8 | 15
  Other | 2 | 2 | 4
  Unknown or Not Reported | 4 | 2 | 6
Annual Household Income [Count of Participants; unit: Participants]
  Less than $40,000 | 11 | 19 | 30
  $40,000-79,999 | 25 | 20 | 45
  $80,000 or More | 22 | 26 | 48
  Unknown or Not Reported | 40 | 35 | 75
Education Level [Count of Participants; unit: Participants]
  High School or Less | 20 | 35 | 55
  Post-high School, but Less than Graduate Degree | 29 | 27 | 56
  Graduate Degree or More | 15 | 11 | 26
  Other | 5 | 6 | 11
  Unknown or Not Reported | 29 | 21 | 50
Parent Clinical Trial [Count of Participants; unit: Participants] — Participants for the ETRIC (BMT CTN 1205) study were recruited from those that were potentially eligible for BMT CTN 0901, 1101, 1203, or 1301 (NCT01339910, NCT01597778, NCT02208037, and NCT02345850, respectively). The parent clinical trial is the BMT CTN trial for which the participant was potentially eligible.
  Participants
    BMT CTN 0901 | 10 | 11 | 21
    BMT CTN 1101 | 25 | 22 | 47
    BMT CTN 1203 | 50 | 51 | 101
    BMT CTN 1301 | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Quality of Informed Consent Part A (QuIC-A) Score
Description: The primary objective of the trial is to compare objective comprehension scores on the Quality of Informed Consent (part A) instrument between subjects randomized to the ETRIC versus the standard consent arms. The QuIC-A is scored on a normalized scale from 0 to 100, with a higher score indicating a greater level of comprehension.
Time Frame: Within 7 days of consent discussion
Population: Participants completing the QuIC-A assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 71 | 81
units on a scale | 81.8 (9.5) | 80.5 (8.7)
Statistical Analysis 1: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in comprehension of the parent clinical trial, as measured by the QuIC-A, between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Mean QuIC-A scores were compared between arms, which should be approximately equal under the null hypothesis; Test type: Superiority; p = 0.37, t-test, 2 sided — Testing was performed at a significance level of 0.05; Two-sample t-test comparing mean QuIC-A scores performed using 150 degrees of freedom

2. Secondary Outcome: Quality of Informed Consent Part B (QuIC-B) Score
Description: The Quality of Informed Consent Part B measures participants' perception of their understanding of cancer clinical trials to address 13 independent domains of informed consent. The QuIC-B is scored on a normalized scale from 0 to 100, with a higher score indicating a greater level of perceived understanding.
Time Frame: Within 7 days of consent discussion
Population: Participants completing the QuIC-B assessment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 71 | 81
units on a scale | 98.2 [91.9 to 100.0] | 96.4 [89.3 to 100.0]
Statistical Analysis 1: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in participants' perception of their comprehension of the parent clinical trial, as measured by the QuIC-B, between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median QuIC-B scores were compared between arms, which should be approximately equal under the null hypothesis; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney) — Testing performed at a significance level of 0.05

3. Secondary Outcome: Modified Deaconess Informed Consent Comprehension Test (DICCT)
Description: The Modified Deaconess Informed Consent Comprehension Test (DICCT) uses semi-structured interviews to assess subject's understanding of the study for which they participated in an informed consent discussion. This modification of the DICCT has 11 items, each scored from 0 to 2 (0 = incorrect, 1 = partially correct, 2 = correct). The item scores are summed to produce a total score ranging from 0 to 22. A higher score indicates a higher level of comprehension.
Time Frame: WIthin 7 days of consent discussion
Population: Participants completing the modified DICCT assessment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 73 | 84
units on a scale | 15 [13 to 17] | 15 [14 to 17]
Statistical Analysis 1: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in participants' comprehension of the parent clinical trial, as measured by the DICCT, between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median DICCT scores were compared between arms, which should be approximately equal under the null hypothesis; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05

4. Secondary Outcome: REALM-R Score
Description: The Rapid Estimate of Adult Literacy in Medicine-Revised (REALM-R) is an 8-item word recognition test to provide clinicians with a valid quick assessment of patient health literacy. The score is computed as the number of words out of 8 that the patient pronounces correctly.
Time Frame: Within 7 days of consent discussion
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 98 | 100
Participants
  Less Than 8 | 15 | 17
  8 | 62 | 69
  Not Completed | 21 | 14

5. Secondary Outcome: Newest Vital Sign (NVS) Score
Description: The Newest Vital Sign is a screening tool that identifies patients at risk for low health literacy. It consists of a nutritional label accompanied by five questions about information on the label. The score is equal to the number of questions answered correctly.
Time Frame: Within 7 days of consent discussion
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 98 | 100
Participants
  Less Than 4 | 11 | 16
  4 | 53 | 52
  5 | 13 | 18
  Not Completed | 21 | 14

6. Secondary Outcome: State Trait Anxiety Inventory (STAI) Score
Description: The State Trait Anxiety Inventory (STAI) measures anxiety and distinguishes it from depressive syndromes. It has two subscales: the State Anxiety Scale evaluates the current state of anxiety, asking how respondents feel "right now," and Trait Anxiety Scale evaluating relatively stable aspects of "anxiety proneness". The STAI has 40 items, 20 items allocated to each subscale, with each item scored on a 4 point Likert scale. The subscale scores shown are averages of the items in the subscale ranging from 1.0 to 4.0, with a higher score indicating a greater level of anxiety.
Time Frame: Within 7 days of consent discussion
Population: Participants completing the STAI assessment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 72 | 80
units on a scale
  State Anxiety Scale | 2.5 [2.3 to 2.6] | 2.5 [2.3 to 2.6]
  Trait Anxiety Scale | 2.4 [2.2 to 2.5] | 2.3 [2.1 to 2.5]
Statistical Analysis 1: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in participants' state anxiety, as measured by the STAI, between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median state anxiety subscores of the STAI were compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in participants' trait anxiety, as measured by the STAI, between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median trait anxiety subscores of the STAI were compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05

7. Secondary Outcome: Participant Satisfaction With Consent Process
Description: A short study specific questionnaire and selected questions from the Quality of Informed Consent (QuIC) supplement questionnaire will query participants about their overall satisfaction with the consent process, helpfulness of information provided, and comprehension of key study-specific elements of treatment. Seven questions are included, each scored on a five point Likert scale. The overall score is the average of the item scores, ranging from 1.0 to 5.0, with a higher score indicating a higher level of satisfaction.
Time Frame: Within 7 days of consent discussion
Population: Participants completing the satisfaction questionnaire
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 72 | 82
units on a scale | 4.2 [3.7 to 4.9] | 4.1 [3.9 to 4.7]
Statistical Analysis 1: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in satisfaction with the consent process, as measured by a study-specific questionnaire, between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median participant satisfaction scores were compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.80, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05

8. Secondary Outcome: Participant Information Location Time
Description: Participants are asked to identify select items within the consent document and the time taken to locate items is measured. Patients who were not able to identify a given section were assigned the maximum time allotted to find each section (180 seconds).
Time Frame: Within 7 days of consent discussion
Population: Participants completing the information location assessment
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 76 | 85
seconds
  Finding Main Goal for Study | 22 [11 to 60] | 30 [11 to 63]
  Finding Who to Contact for Questions | 15 [7 to 34] | 20 [10 to 45]
  Finding Risks and Benefits Section | 20 [14 to 30] | 20 [10 to 40]
  Finding How to Leave the Study | 24 [15 to 60] | 30 [11 to 60]
  Finding Study Procedures | 43 [21 to 83] | 36 [18 to 96]
Statistical Analysis 1: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the time required to find the main goal of the study between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median time required to find the main goal of the study was compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the time required to find who to contact for questions between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median time required to find who to contact for questions was compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05
Statistical Analysis 3: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the time required to find the risks and benefits section between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median time required to find the risks and benefits section was compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05
Statistical Analysis 4: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the time required to find how to leave the study between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median time required to find how to leave the study was compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05
Statistical Analysis 5: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the time required to find study procedures between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Median time required to find study procedures was compared between arms, which should be equal under the null hypothesis; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney) — Testing was performed at a significance level of 0.05

9. Secondary Outcome: Consent Rate on Parent Trial
Description: The consent rate is the rate at which participants provided consent to participate in the parent trial.
Time Frame: Within 7 days of consent discussion
Population: Consent rates are computed specific to each trial
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Number analyzed (Participants) | 98 | 100
Participants
  BMT CTN 0901: number analyzed (Participants) | 10 | 11
  BMT CTN 0901 | 2 | 3
  BMT CTN 1101: number analyzed (Participants) | 25 | 22
  BMT CTN 1101 | 13 | 10
  BMT CTN 1203: number analyzed (Participants) | 50 | 51
  BMT CTN 1203 | 22 | 25
  BMT CTN 1501: number analyzed (Participants) | 13 | 16
  BMT CTN 1501 | 9 | 7
Statistical Analysis 1: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the consent rates to BMT CTN 0901 between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Consent rates to BMT CTN 0901 were compared between arms in participants considering enrollment, which should be equal under the null hypothesis; Test type: Superiority; p = 1.00, Fisher Exact — Testing was performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the consent rates to BMT CTN 1101 between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Consent rates to BMT CTN 1101 were compared between arms in participants considering enrollment, which should be approximately equal under the null hypothesis; Test type: Superiority; p = 0.77, Fisher Exact — Testing was performed at a significance level of 0.05
Statistical Analysis 3: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the consent rates to BMT CTN 1203 between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Consent rates to BMT CTN 1203 were compared between arms in participants considering enrollment, which should be approximately equal under the null hypothesis; Test type: Superiority; p = 0.69, Fisher Exact — Testing was performed at a significance level of 0.05
Statistical Analysis 4: Comparison: Standard Consent vs Easy-to-Read Informed Consent; The null hypothesis is that there is no difference in the consent rates to BMT CTN 1301 between participants reviewing a standard consent and easy-to-read informed consent (ETRIC) forms. Consent rates to BMT CTN 1501 were compared between arms in participants considering enrollment, which should be approximately equal under the null hypothesis; Test type: Superiority; p = 0.26, Fisher Exact — Testing was performed at a significance level of 0.05

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not monitored.
Arm/Group | Standard Consent | Easy-to-Read Informed Consent
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT02081248/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2016-09-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT02081248/SAP_001.pdf